CLINICAL TRIAL: NCT05000710
Title: Single Arm Phase II, Multicenter Study of Concomitant Radiotherapy, Tremelimumab and Durvalumab (MEDI4736) for Metastatic or Locally Advanced NSCLC Patients Progressing on First-line Immunotherapy
Brief Title: Concomitant Radiotherapy, Tremelimumab & Durvalumab for Advanced NSCLC Patients Progressing on First-line Immunotherapy
Acronym: CORAL-Lung
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: AstraZeneca (Industry); Rambam Health Care Campus (Other); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Jair Bar, M.D., Ph.D., Deputy Director, Institute of Oncology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-17-13252
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Metastatic or Locally Advanced NSCLC
Keywords: checkpoint inhibitors; treatment-related toxicity leading to treatment discontinuation; RECIST 1.1
MeSH Terms: conditions — Neoplasm Metastasis | interventions — durvalumab; tremelimumab; Radiation

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study arm (Experimental): Study treatments include:
  Durvalumab at D1 and q4w + Tremelimumab at C1D1 and C4D1. Radiotherapy 11 fractions (start at D21).
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Low dose irradiation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab administered IV over 60 minutes at a dose of 1500 mg every 4 weeks
  Other Names: Imfinzi; MEDI4736
Drug: Tremelimumab — Tremelimumab administered IV over 60 minutes at a dose of 300 mg , twice: at C1D1 and C4D1
Radiation: Low dose irradiation — 21 days after the first immunotherapy treatment 11 fractions of 3 Gy will be administrated to metastatic or primary lesion/s over 2 weeks and one day

SUMMARY:
This is an open-label, single-arm, phase 2a trial with a safety run-in cohort followed by a Simon two-step design expansion cohort, of two checkpoint blockage treatments and radiotherapy in the treatment of locally advanced or metastatic NSCLC who have failed first-line immunotherapy (alone or as a combination regimen with chemotherapy).

Study objectives:

Objective of the safety run-in phase:

• To evaluate safety of the triple combination of irradiation -Durvalumab - Tremelimumab

Co-Primary objectives of the entire study:

* To evaluate safety of the triple combination (as for the run-in phase).
* To evaluate response rate on study drug compared to historical data of response to first-line platinum-doublet chemotherapy and 2nd-line docetaxel.

Secondary objective:

• To evaluate PFS and OS compared to historical data .

Exploratory objectives:

* Examine the mechanism of resistance to first-line immunotherapy .
* Examine the immune response in irradiation -Durvalumab - Tremelimumab treated patients and identify potential predictors of clinical benefit.

DETAILED DESCRIPTION:
A cycle is defined as 28 days. Eligible patients who have a radiologically confirmed progressive disease on first line Immunotherapy treatment will receive an intravenous injection of 300 mg Tremelimumab at D1 and 12 weeks later a second dose of 300 mg tremelimumab, and an intravenous injections of 1500 mg Durvalumab q4w (starting from D1) . Treatment duration is until objective radiological disease progression as per RECIST 1.1 assessed by the local radiologist, and as long as the patients are benefiting from treatment according to the investigator's opinion and they do not meet any other discontinuation criteria.

21 days after the first immunotherapy treatment, a radiotherapy course of 11 fractions of 3 Gy (total of 33 Gy) will be administrated to metastatic or primary lesion/s over two weeks and one day. The second durvalumab treatment will be administered at the beginning of the 2nd week of radiotherapy, one week after radiotherapy start day.

Following patients consent, a fresh biopsy specimen will be obtained (if not previously obtained after PD) for correlative studies, preferably from site of disease progression on first line immunotherapy.

In addition, tissue samples will be obtained from both existing archived biopsy (diagnostic specimen), if available. An optional newly biopsied tissue sample will be taken 20 weeks after initiation of study treatment and at the time of progression on study treatment. Biopsy at PD is mandatory if can be performed with no significant risk.

Blood and microbiome samples for correlative studies will be taken at predefined intervals, to explore predictive biomarkers for clinical efficacy, determine pharmacodynamic effects on immune cells, determine immune response signatures.

Tumor imaging should be acquired by CT and include the chest, abdomen, and pelvis with and without IV contrast and with oral contrast. CT should be performed at baseline and every 8 weeks until objective radiological disease progression assessed as per RECIST 1.1.

Patients who have discontinued treatment should be seen at end of treatment and 28 days post discontinuation for the evaluations outlined in the study schedule. Patients will be contacted every 90 days following discontinuation visit to capture survival status.

Any patient who discontinues study treatment for reasons other than objective radiological progression should continue to undergo scheduled objective tumor assessments according to the study schedule in order to assess objective radiological progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic (stage 3 or stage 4) histologically proven NSCLC patients not candidate for curative - intent treatment.
* Have been previously treated with one prior immunotherapy (i.e. anti-PD1 or anti-PD-L1 antibodies, with or without chemotherapy) for advanced or metastatic NSCLC. Additional systemic treatment lines for metastatic disease are not allowed.

  1. Previous chemotherapy treatment lines administered earlier for non-metastatic disease (adjuvant, neo-adjuvant) are allowed if completed more than six months prior to diagnosis of advanced disease.
  2. Patients recurring within six months of end of adjuvant/maintenance immunotherapy (e.g. durvalumab post-chemorads) are eligible for the study if no additional systemic treatment was administered prior to enrollment on the study (this situation is considered equivalent to progression on first-line immunotherapy).
* Documented radiologic progression on immunotherapy. Minimal treatment time on first-line immunotherapy is 12 weeks. Progressive disease needs to be confirmed by a repeat scan performed at least 4 weeks after the first objective progression.
* Availability of at least 1 disease site not previously irradiated to serve as a target for radiotherapy. However, a disease site that progressed after having received previously radiotherapy can serve as a radiotherapy target on this trial.
* Availability of at least 1 measurable lesion not previously irradiated that is not planned to be irradiated during the study and measurable as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Availability of at least 1 disease site suitable for biopsy procedure (unless the patient has had a biopsy postprogression on immunotherapy), preferably, at site of disease progression on immunotherapy. Fine needle aspirate , ascites or effusion specimens are not acceptable . Selected sites for biopsy can serve afterwards as radiotherapy targets.
* Patient must have had a treatment free interval of at least 4 weeks from any prior therapy (includes major surgery) before starting of study drugs.

Minor surgical procedures (as defined by the investigator): 7 post-operative days.

Patients who receive palliative radiation for nontarget tumour lesions need a washout period of 7 days.

* Have an ECOG performance status of 0 or 1 and a minimum life expectancy of 12 weeks.
* Have adequate normal organ and marrow function, including the following:

  1. Absolute neutrophil count ≥1.0 × 109/L.
  2. Platelet count ≥ 75× 109/L.
  3. Haemoglobin ≥ 9.0 g/dL.
  4. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 × the upper limit of normal (ULN) if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
  5. Total bilirubin (TBL) ≤ 1.5 × ULN or for patients with documented/suspected Gilbert's disease, bilirubin ≤ 2 × ULN.
  6. Creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 40 mL/min (creatinine clearance can be measured or calculated by Cockcroft and Gault equation; measurement/calculation is only required when creatinine is >1.5 × ULN).
* Body weight >30kg
* Be willing and able to provide written informed consent for the trial prior to any study specific procedures.The subject must also provide consent for correlative translational study.
* Male or female subjects who are ≥ 18 years of age on the day of signing the informed consent.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of study medication.
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 180 days after the last dose of study therapy.

Exclusion Criteria:

* Progression (as defined by RECIST 1.1) within 12 weeks from initiation of immunotherapy (this criteria aims at exclusion of patients with primary resistance; this study focuses on acquired resistance).
* Prior exposure to anti CTLA-4, including tremelimumab
* All potential radiotherapy targets involve high risk of significant toxicity.
* Mixed response to immunotherapy, where growth occurred only in a single lesion that is amendable to curative-intent radiotherapy (this criteria aims to exclude patients more likely to benefit from targeted radiotherapy to the growing mass and continuation of immunotherapy).
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Any prior immune-related adverse events grade 3 or higher (as per CTCAE version 5.0).
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Progressing brain metastasis. Stable brain metastasis (based on at least two brain imaging tests with a 4 week interval or more) are allowed (including non-treated lesions) as long as there no requirement for steroids due to the brain spread for ≥4 weeks prior to start of study treatment.
* History of leptomeningeal carcinomatosis
* Patients whose tumour samples are known to have activating mutations in the EGFR gene, translocations of the ALK gene, or rearrangement of the ROS1 gene that are indicated for treatment by approved TKI therapy are excluded.
* Autoimmune or inflammatory disorders requiring systemic treatment during the year prior to study treatment including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, celiac disease (or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis. The following are exceptions to this criterion: Patients with vitiglio or alopecia, Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable on hormone replacement not requiring systemic treatment, Psoriasis not requiring treatment. Additional exceptions are any chronic skin condition that does not require systemic therapy and patients with celiac disease controlled by diet alone. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion: Intranasal, inhaled, or topical steroids, or local steroid injections (e.g., intraarticular injection). Systemic corticosteroids at physiologic doses are allowed up to 10 mg/day of prednisone or its equivalent. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) are allowed.
* Active infection with hepatitis B (known positive HBV surface antigen[HBsAg] result), hepatitis C or tuberculosis. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg are eligible.Patients positive for hepatitis C (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV RNA. Tuberculosis clinical evaluation includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice.
* Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
* Organ transplanted patients.
* Any condition that, in the opinion of the Investigator, would interfere with the evaluation of IP or interpretation of patient safety or study results, including, but not limited to, uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of another primary malignancy except for: Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IP and of low potential risk for recurrence, Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated carcinoma in situ (breast DCIS, non-invasive cervical cancer, etc.) without evidence of disease. Patients with tumors with a very low risk of metastatic spread and recurrence that were treated successfully with a curative intent (e.g. resected local carcinoid tumor, recected low grade, non-muscle invasive bladder cancer) can be considered for inclusion based on decision of the study physician.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drugs.
* Have received treatment with an investigational product or nonapproved use of a drug or device within 28 days prior to the initial dose of study drugs, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Female patients who are pregnant or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
treatment-related toxicity leading to treatment discontinuation (TRTLTD), as assessed by CTC-AE version 5.0. | Approximately 2 years
  number of patients with TRTLTD will be evaluated during the safety run-in phase
Incidence of Treatment-Emergent Adverse Events, as assessed by CTCAE version 5.0 | From day of subject's written consent until study termination, approximately 4.5 years
  Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, most updated version) terminology and presented in tables by System Organ Class (SOC) and Preferred Term (PT).
Response rate on study treatment (according to investigator assessment, per RECIST 1.1) | Up to 5 months from treatment initiation, approximately 4.5 years overall
  Proportion of subjects showing best overall response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
PFS on study treatment (according to investigator assessement, per RECIST 1.1 | From first dose of immunotherapy until first progression, approximately 4.5 years
  Duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | From documented metastatic disease until death (or date of last documentation of being alive), approximately 4.5 years
  Duration of time from diagnosis until death (or date of last documentation of being alive). Survival data may be obtained via contact with the patient, patient's family, or through a review of the patient's notes, or through the use of public records.
Change in biomarkers | 5 years
  Blood, tumor and microbiome samples will be analyzed for various biomarkers. Initial biomarkers to be tested include proteins such as PDL-1, immune cell composition, cfDNA, microRNA proteomics and bacteria populations

CONTACTS AND LOCATIONS:
Overall Officials: Jair Bar, Dr, Principal Investigator — Shaba Medical Center
Locations (1):
- Sheba Medical Centre, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frey B, Ruckert M, Weber J, Mayr X, Derer A, Lotter M, Bert C, Rodel F, Fietkau R, Gaipl US. Hypofractionated Irradiation Has Immune Stimulatory Potential and Induces a Timely Restricted Infiltration of Immune Cells in Colon Cancer Tumors. Front Immunol. 2017 Mar 8;8:231. doi: 10.3389/fimmu.2017.00231. eCollection 2017. PMID 28337197
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Klug F, Prakash H, Huber PE, Seibel T, Bender N, Halama N, Pfirschke C, Voss RH, Timke C, Umansky L, Klapproth K, Schakel K, Garbi N, Jager D, Weitz J, Schmitz-Winnenthal H, Hammerling GJ, Beckhove P. Low-dose irradiation programs macrophage differentiation to an iNOS(+)/M1 phenotype that orchestrates effective T cell immunotherapy. Cancer Cell. 2013 Nov 11;24(5):589-602. doi: 10.1016/j.ccr.2013.09.014. Epub 2013 Oct 24. PMID 24209604
- [Background] Chajon E, Castelli J, Marsiglia H, De Crevoisier R. The synergistic effect of radiotherapy and immunotherapy: A promising but not simple partnership. Crit Rev Oncol Hematol. 2017 Mar;111:124-132. doi: 10.1016/j.critrevonc.2017.01.017. Epub 2017 Feb 4. PMID 28259287
- [Background] McNamara MJ, Hilgart-Martiszus I, Barragan Echenique DM, Linch SN, Kasiewicz MJ, Redmond WL. Interferon-gamma Production by Peripheral Lymphocytes Predicts Survival of Tumor-Bearing Mice Receiving Dual PD-1/CTLA-4 Blockade. Cancer Immunol Res. 2016 Aug;4(8):650-7. doi: 10.1158/2326-6066.CIR-16-0022. Epub 2016 Jun 4. PMID 27262113
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610